CLINICAL TRIAL: NCT04302714
Title: Hysteroscopic vs. Cervical Injection for Sentinel Node Detection of Endometrial Cancer: a Multicenter Prospective Randomized Study
Brief Title: Hysteroscopic vs. Cervical Injection for Sentinel Node Detection of Endometrial Cancer
Acronym: SLN_EC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 09/17
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Cancer
Keywords: Cervical injection; Hysteroscopic injection
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical injection (Active Comparator): Fluorescent SLN Imaging With Indocyanine Green (ICG), using near-infrared fluorescence imaging, will be used as a dye for SLN mapping. Injections will be performed intraoperative. Concentration of ICG used is 1.25mg/mL, the 25mg dry powder bottle is mixed with 20 mL of sterile water in the operating room, and 4 mL is injected directly into the cervix. This solution was injected intracervically at 3 and 9 o'clock positions, both submucosally and deep into the cervical stroma. A spinal needle 18-gauce is used to inject the ICG. The 4 mL can be divided into 4 separate injections (1 mL each). The ICG should be injected slowly, at a rate of 5 to 10 seconds per quadrant.
  Interventions: Procedure: Cervical injection
- hysteroscopic injection (Experimental): hysteroscopy is performed using an operative hysteroscope. Uterine distension is obtained by means of saline solution. Usually, the fluid bag is placed 50 cm above the patient's plane so that the intracavitary pressure does not exceed 40 mm Hg. After visualization of uterine cavity a 22-gauce, 40-mm needle was introduced into the operative port and IGC is injected peritumorally. Concentration of ICG used is 1.25mg/mL, the 25mg dry powder bottle is mixed with 20 mL of sterile water in the operating room. The injection is performed subendometrially around the lesion, or, if the uterine cavity was totally involved by disease, at 3, 6, 9, and 12 o'clock . The depth of needle placement is modulated by visualizing endometrial elevation during injection.
  Interventions: Procedure: Hysteroscopic injection

INTERVENTIONS:
Procedure: Hysteroscopic injection — Hysteroscopic injection
  Arms: hysteroscopic injection
Procedure: Cervical injection — Cervical injection
  Arms: cervical injection

SUMMARY:
Hysteroscopic vs. Cervical Injection for Sentinel Node Detection of Endometrial Cancer: a multicenter prospective randomized study

DETAILED DESCRIPTION:
Hysteroscopic vs. Cervical Injection for Sentinel Node Detection of Endometrial Cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from the patient;
* Histological diagnosis of endometrial cancer (including type I and II EC);
* Early stage (FIGO stage < 4);
* Age older than 18 years.

Exclusion Criteria:

* Preoperative diagnosis of extra-uterine disease;
* Preoperative suspicious of gross positive nodes;
* Execution of neoadjuvant chemotherapy;
* Contraindication to upfront general anesthesia and or mini-invasive surgery;
* Systemic infections ongoing;
* Pregnancy ongoing.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Detection rate | 30 month
  assessment of Detection rate in the para-aortic area

SECONDARY OUTCOMES:
Detection rate | 30 month
  Detection rate in the pelvic area
Operative time | 30 month
  Operative time to detect and remove sentinel node
Intraoperative complications | 30 month
  Intraoperative complications during the sentinel lymph node dissection
Postoperative complications | 30 month
  Postoperative complications graded per the Clavien-Dindo Classification system

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Ditto, MD, Principal Investigator — Fonsazione IRCCS Istituto Nazionale Tumori Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

REFERENCES:
- [Background] Martinelli F, Ditto A, Bogani G, Signorelli M, Chiappa V, Lorusso D, Haeusler E, Raspagliesi F. Laparoscopic Sentinel Node Mapping in Endometrial Cancer After Hysteroscopic Injection of Indocyanine Green. J Minim Invasive Gynecol. 2017 Jan 1;24(1):89-93. doi: 10.1016/j.jmig.2016.09.020. Epub 2016 Oct 8. PMID 27725278
- [Background] Maccauro M, Lucignani G, Aliberti G, Villano C, Castellani MR, Solima E, Bombardieri E. Sentinel lymph node detection following the hysteroscopic peritumoural injection of 99mTc-labelled albumin nanocolloid in endometrial cancer. Eur J Nucl Med Mol Imaging. 2005 May;32(5):569-74. doi: 10.1007/s00259-004-1709-4. Epub 2004 Dec 30. PMID 15625604
- [Background] Raspagliesi F, Ditto A, Kusamura S, Fontanelli R, Vecchione F, Maccauro M, Solima E. Hysteroscopic injection of tracers in sentinel node detection of endometrial cancer: a feasibility study. Am J Obstet Gynecol. 2004 Aug;191(2):435-9. doi: 10.1016/j.ajog.2004.03.008. PMID 15343218
- [Background] Niikura H, Okamura C, Utsunomiya H, Yoshinaga K, Akahira J, Ito K, Yaegashi N. Sentinel lymph node detection in patients with endometrial cancer. Gynecol Oncol. 2004 Feb;92(2):669-74. doi: 10.1016/j.ygyno.2003.10.039. PMID 14766264
- [Background] Gargiulo T, Giusti M, Bottero A, Leo L, Brokaj L, Armellino F, Palladin L. Sentinel Lymph Node (SLN) laparoscopic assessment early stage in endometrial cancer. Minerva Ginecol. 2003 Jun;55(3):259-62. PMID 14581872
- [Background] Pelosi E, Arena V, Baudino B, Bello M, Giusti M, Gargiulo T, Palladin D, Bisi G. Pre-operative lymphatic mapping and intra-operative sentinel lymph node detection in early stage endometrial cancer. Nucl Med Commun. 2003 Sep;24(9):971-5. doi: 10.1097/00006231-200309000-00005. PMID 12960596
- [Background] Pelosi E, Arena V, Baudino B, Bello M, Gargiulo T, Giusti M, Bottero A, Leo L, Armellino F, Palladin D, Bisi G. Preliminary study of sentinel node identification with 99mTc colloid and blue dye in patients with endometrial cancer. Tumori. 2002 May-Jun;88(3):S9-10. doi: 10.1177/030089160208800322. PMID 12365393
- [Background] Ditto A, Martinelli F, Bogani G, Papadia A, Lorusso D, Raspagliesi F. Sentinel node mapping using hysteroscopic injection of indocyanine green and laparoscopic near-infrared fluorescence imaging in endometrial cancer staging. J Minim Invasive Gynecol. 2015 Jan;22(1):132-3. doi: 10.1016/j.jmig.2014.08.009. Epub 2014 Aug 15. PMID 25135786
- [Background] Solima E, Martinelli F, Ditto A, Maccauro M, Carcangiu M, Mariani L, Kusamura S, Fontanelli R, Grijuela B, Raspagliesi F. Diagnostic accuracy of sentinel node in endometrial cancer by using hysteroscopic injection of radiolabeled tracer. Gynecol Oncol. 2012 Sep;126(3):419-23. doi: 10.1016/j.ygyno.2012.05.025. Epub 2012 May 30. PMID 22659192
- [Background] Perrone AM, Casadio P, Formelli G, Levorato M, Ghi T, Costa S, Meriggiola MC, Pelusi G. Cervical and hysteroscopic injection for identification of sentinel lymph node in endometrial cancer. Gynecol Oncol. 2008 Oct;111(1):62-7. doi: 10.1016/j.ygyno.2008.05.032. Epub 2008 Jul 14. PMID 18625518
- [Background] Cormier B, Rozenholc AT, Gotlieb W, Plante M, Giede C; Communities of Practice (CoP) Group of Society of Gynecologic Oncology of Canada (GOC). Sentinel lymph node procedure in endometrial cancer: A systematic review and proposal for standardization of future research. Gynecol Oncol. 2015 Aug;138(2):478-85. doi: 10.1016/j.ygyno.2015.05.039. Epub 2015 Jun 3. PMID 26047592